CLINICAL TRIAL: NCT01549769
Title: A Multiple-Dose, Open-Label Pharmakokinetic and Pharmacodynamic Study of Bardoxolone Methyl in Patients With Chronic Kidney Disease and Type 2 Diabetes
Brief Title: Pharmacokinetic and Pharmacodynamic Study of Bardoxolone Methyl in Patients With Chronic Kidney Disease and Type 2 Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: IDMC recommendation for safety concerns
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-1102
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — bardoxolone methyl

ARMS (1):
- Bardoxolone Methyl 20 mg (Experimental)
  Interventions: Drug: Bardoxolone Methyl

INTERVENTIONS:
Drug: Bardoxolone Methyl — Oral, once daily

SUMMARY:
This study is to evaluate the pharmacokinetics and pharmacodynamics of bardoxolone methyl in patients with chronic kidney disease and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Screening eGFR ≥ 15.0 and < 45.0 mL/min/1.73 m2.
2. A history of type 2 diabetes; diagnosis should have been made at ≥ 30 years of age (if diabetes developed at a younger age, a fasting C-peptide level must confirm type 2 diabetes);
3. Male or female patients at least 18 years of age;
4. Body mass index (BMI) between 18.5 and 45 kg/m2;
5. Treatment with an angiotensin converting enzyme (ACE) inhibitor and/or an angiotensin II receptor blocker (ARB) for at least 6 weeks prior to Study Day -1. The dosage of ACE inhibitor and/or ARB must be stable for 2 weeks prior to Screening (i.e., no change in dosage or medication). Patients not taking an ACE inhibitor and/or ARB, or taking an ACE inhibitor and/or ARB at levels below the goal dose set by K/DOQI guidelines (see Appendix B) must have a documented medical contraindication (e.g., hyperkalemia, hypotension), which the investigator must provide and discuss with a medical monitor prior to Study Day -1. Patients not taking an ACE inhibitor and/or ARB because of a medical contraindication must have discontinued treatment at least 8 weeks prior to Screening;
6. Mean systolic blood pressure (SBP) must be ≤ 160 mmHg and ≥ 105 mmHg and mean diastolic blood pressure (DBP) must be ≤ 90 mmHg during screening;
7. Willing to practice methods of birth control (both males who have partners of childbearing potential and females of childbearing potential) from screening through Study Day 84;
8. Female patients of childbearing potential must be non-pregnant and non-lactating and have a negative serum pregnancy test result prior to enrollment in the study;
9. Willing and able to give written informed consent for study participation;
10. Willing and able to cooperate with all aspects of the protocol;

Exclusion Criteria:

1. Type 1 diabetes mellitus (juvenile onset). If a history of diabetic ketoacidosis exists, a fasting C-peptide level must confirm type 2 diabetes;
2. History of a renal transplant or a planned transplant from a living donor during the study;
3. Hemoglobin A1c level > 11.0% (97 mmol/mol) during screening;
4. Acute dialysis or acute kidney injury within 24 weeks prior to Study Day -1;
5. Clinical signs and/or symptoms of uremia and expected need for renal replacement therapy within 12 weeks following Study Day -1, as assessed by the investigator;
6. Albumin/creatinine ratio (ACR) > 3500 mg/g during screening;
7. Recently active cardiovascular disease defined as:

   * Unstable angina pectoris within 12 weeks before Study Day -1;
   * Myocardial infarction, coronary artery bypass graft surgery, or percutaneous transluminal coronary angioplasty/stent within 12 weeks before Study Day -1;
   * Cerebrovascular accident, including transient ischemic attack within 12 weeks before Study Day -1;
   * Current diagnosis of Class III or IV NYHA congestive heart failure (Appendix C);
8. Clinical diagnosis of severe obstructive valvular heart disease or severe obstructive hypertrophic cardiomyopathy;
9. Atrioventricular block, 2° or 3°, not successfully treated with a pacemaker;
10. Diagnostic or interventional procedure that required a contrast agent that may induce nephropathy within 30 days prior to Study Day -1, or planned during the study;
11. Systemic immunosuppression for more than 15 days , cumulatively, within the 12 weeks prior to Study Day -1, or anticipated need for immunosuppression during the study;
12. Total bilirubin, aspartate transaminase (AST), or alanine transaminase (ALT) level greater than the upper limit of normal (ULN) or alkaline phosphatase level greater than two times the ULN on ANY screening laboratory test result;
13. Iron saturation < 20% on Study Day -1. If iron saturation is < 20% at screening, iron supplements may be provided prior to Study Day -3;
14. Serum magnesium levels < 1.3 mEg/L (0.65 mmol/L) on Study Day -1. If serum magnesium levels are < 1.3 mEg/L (0.65 mmol/L) at screening, oral magnesium replacement may be provided prior to Study Day -3;
15. Known hypersensitivity to any component of the study drug;
16. Current history of drug or alcohol abuse, as assessed by the investigator;
17. Clinically significant infection requiring intravenous administration of antibiotics or hospitalization within 6 weeks prior to Study Day -1;
18. Donation or receipt of blood or blood components within the 4 weeks prior to Study Day -1. The investigator should instruct patients who participate in this study not to donate blood or blood components for 4 weeks after the completion of the study;
19. Abnormal ECG at screening, which is interpreted by the investigator to be clinically significant;
20. Use of tobacco-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, etc.) or products for smoking cessation 2 weeks prior to Study Day -1;
21. Treated with any investigational agent within 30 days before Study Day -1, 5 half-lives, or twice the duration of biological effect of the previous investigational drug (whichever is longer);
22. A clinical condition that, in the judgment of the investigator, could potentially pose a health risk to the patient while involved in the study;
23. Participation in a clinical study involving any intervention within 30 days prior to Study Day -1, concurrent participation in such a study, or participation in a prior clinical study involving bardoxolone methyl in any form;
24. Unable to communicate or cooperate with the investigator due to language problems, poor mental development or impaired cerebral function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2012-11-30 (Actual); Study Completion 2013-10-31 (Actual)

PRIMARY OUTCOMES:
Area under the curve | 24 hours

SECONDARY OUTCOMES:
Time to maximum observed concentration | 56 days
Area under the plasma concentration-time curve | 0 to last observed concentration
Maximum observed concentration | 56 days

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/